CLINICAL TRIAL: NCT00958841
Title: An Open Label, Multicenter, Single Arm Study of Pasireotide LAR in Patients With Rare Tumors of Neuroendocrine Origin
Brief Title: Study of Pasireotide in Patients With Rare Tumors of Neuroendocrine Origin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment rate into this study with rare tumors of neuroendocrine origin (enrollment issues)
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230D2203; 2008-007348-32 (EudraCT Number)
Record Dates: First submitted 2009-07-22; First posted 2009-08-13 (Estimated); Results first posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-06

CONDITIONS: Pancreatic Neoplasm; Pituitary Neoplasm; Nelson Syndrome; Ectopic ACTH Syndrome
Keywords: Rare tumors of neuroendocrine origin; NETs of the pancreatic; Pituitary NETs; EAS Tumors; Nelson's Syndrome; Pancreatic neoplasm; pituitary neoplasm; Nelson Syndrome; ectopic ACTH syndrome; pasireotide LAR; PNETs; PiNETS
MeSH Terms: conditions — Pancreatic Neoplasms; Pituitary Neoplasms; Nelson Syndrome; ACTH Syndrome, Ectopic; Neuroectodermal Tumors, Primitive | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pasireotide LAR 60mg (Experimental): Patients received pasireotide LAR at 60 mg approximately once every 28 days for 6 months during the core treatment period and additional treatment cycles up to a total of 48 months during the extension phase.
  Interventions: Drug: pasireotide LAR

INTERVENTIONS:
Drug: pasireotide LAR — Investigational drug pasireotide LAR was supplied in vials with 20 mg or 40 mg powder and 2 mL vehicle was supplied in ampoules for reconstitution.
  Other Names: SOM230

SUMMARY:
This study will assess the effectiveness and safety of pasireotide long-acting release in patients who have rare tumors of neuroendocrine origin.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Patients at least 18 years old
* Patient who have rare tumors of neuroendocrine origin, such as tumors of the:

  1. pancreas
  2. pituitary glands
  3. Nelson syndrome
  4. ectopic-ACTH secreting tumor
* Patients who have failed standard of care treatment or for whom no standard of care treatment exist
* Signed Informed Consent

Exclusion Criteria:

* Patients with active gallbladder disease
* Patients with any ongoing or planned anti-neoplastic or interferon therapy
* Poorly controlled diabetes mellitus
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (39):
- United States (6):
  - Cedars Sinai Medical Center Cedars Sinai 4, Los Angeles, California
  - Cedars Sinai Medical Center The Pituitary Center (3), Los Angeles, California
  - Stanford University Medical Center SC, Stanford, California
  - Dana Farber Cancer Institute Deptof DanaFarberCancerInst(5), Boston, Massachusetts
  - Mount Sinai School of Medicine Study Coordinator, New York, New York
  - Swedish Medical Center Dept.ofSwedishMedicalCtr.(2), Seattle, Washington
- Novartis Investigative Site, Buenos Aires, Buenos Aires, Argentina
- Australia (2):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Fitzroy, Victoria
- Brazil (3):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Botucatu, São Paulo
- Canada (2):
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Montreal, Quebec
- France (8):
  - Novartis Investigative Site, Strasbourg, France
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Reims
- Germany (6):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg
- Italy (5):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Mexico City, Mexico City, Mexico
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (2):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
- Novartis Investigative Site, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For all other individual indications, the numbers of patients in the efficacy analyzable sets were less than 6 and therefore no responder analyses were carried out for these indications.
Groups:
- Pasireotide LAR 60mg: All patients received pasireotide LAR at 60 mg approximately once every 28 days for 6 months during the core treatment period and additional treatment cycles up to a total of 48 months during the extension phase. Patients included patients with pancreatic neuroendocrine tumors (PNETs), pituitary NETs (PiNETs), Ectopic ACTH-secreting tumor (EAS) & Nelson's syndrome.
Period: Overall Study
Arm/Group | Pasireotide LAR 60mg
Started | 118
Completed Month 6 (M6) | 90
Entered in Extension | 63
Completed | 22 (Completed = Completed extension)
Not Completed | 96
Not completed — Abnormal laboratory value(s) | 1
Not completed — Abnormal test procedure result(s) | 3
Not completed — Administrative problems | 1
Not completed — Adverse Event | 8
Not completed — New cancer therapy | 5
Not completed — Withdrawal by Subject | 1
Not completed — Unsatisfactory therapeutic effect | 22
Not completed — Completed M6/did not enter extension | 27
Not completed — Discontinued prior to M* | 28

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all enrolled patients who received at least one dose of pasireotide LAR.
Arm/Group | Pasireotide LAR 60mg
Number analyzed (Participants) | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (14.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders at Month 6 - Pooled Pancreatic NETs (PNETs)
Description: The primary efficacy endpoint was defined as the percentage of responders at Month 6 among pooled PNET patients (insulinoma, gastrinoma, VIPoma, and glucagonoma). A responder was defined as a patient who either attained normalization or had a greater than 50% reduction from baseline of the level of the primary biochemical tumor marker at Month 6 (M6). Four insulinoma pts were excluded from analysis because of unavailability of normal ranges for the associated primary biochemical tumor marker (insulin-to-glucose ratio). One patient with VIPoma with a normal baseline was also excluded. As a result, only 20 out of 25 patients with PNET were included in the assessment of the primary endpoint, which was less than the planned sample size of 34. Therefore, the primary objective could not be assessed with sufficient power. Patients with missing Month 6 assessment were considered as non-responders. Responder analyses are reported only for indications with minimum of 6 patients.
Time Frame: 6 months
Population: The efficacy analyzable set included all enrolled patients who received at least one dose of pasireotide LAR and had indication-specific baseline primary biochemical tumor marker levels >ULN. Patients with baseline primary biochemical tumor marker levels either missing at baseline or missing ULN or baseline value ≤ ULN were excluded.
Measure: Number; unit: percentage of participants
Groups:
- Gastrinoma; VIpoma; Glucagonoma: One of the 10 types of PNETs analyzed
Arm/Group | Gastrinoma | VIpoma | Glucagonoma
Number analyzed (Participants) | 13 | 2 | 5
percentage of participants | 46.2 | 0.0 | 0.0

2. Secondary Outcome: Percentage of Responders at Month 6 - Individual NETs
Description: Percentage of responders for each of the 10 NET indications considered in the study. Responder analyses were performed for an indication only if there were at least 6 patients in the efficacy analyzable set. For all other individual indications, the numbers of patients in the efficacy analyzable sets were less than 6 and therefore no responder analyses were carried out for these indications.
Time Frame: 6 months
Population: The efficacy analyzable set included all enrolled patients who received at least one dose of pasireotide LAR and had indication-specific baseline primary biochemical tumor marker levels >ULN.
Measure: Number; unit: percentage of participants
Groups:
- Prolactinoma: One of the 10 types of PNETs analyzed.
- Nelson's Syndrome: based on disease specific primary biochemical tumor markers. Patients received pasireotide LAR at 60 mg approximately once every 28 days for 6 months during the core treatment period and additional treatment cycles up to a total of 48 months during the extension phase.
Arm/Group | Gastrinoma | Prolactinoma | Nelson's Syndrome
Number analyzed (Participants) | 13 | 37 | 14
percentage of participants | 46.2 | 21.6 | 50.0

3. Secondary Outcome: Percentage of Responders With Probability of Success at Month 6 - Individual NETs
Description: Percentage of responders for each of the 10 NET indications considered in the study. Responder analyses were performed for an indication only if there were at least 6 patients in the efficacy analyzable set. For all other individual indications, the numbers of patients in the efficacy analyzable sets were less than 6 and therefore no responder analyses were carried out for these indications. The probability of success was a chance that the true responder rate was greater than 15%) for the indications gastrinoma, prolactinoma, and Nelson's syndrome.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Gastrinoma | Prolactinoma | Nelson's Syndrome
Number analyzed (Participants) | 13 | 37 | 14
Percentage of participants | 46.2 | 21.6 | 50.0

4. Secondary Outcome: PNETs: Number of Patients Attaining Normalization or a More Than 50% Reduction in Primary Biochemical Tumor Marker
Description: Specific primary biochemical tumor markers were used to assess the efficacy of pasireotide in PNETs. A Month 6 responder was defined as the patients who either attained normalization or greater than 50% reduction from baseline in the level of the primary biochemical tumor marker at Month 6. One gastrinoma patient had a missing primary tumor marker value at Month 6, but had a Month 5 assessment done on Day 141, which fell within the allowed window period for Month 6.
Time Frame: Baseline, month 6
Population: The efficacy analyzable set included all enrolled patients who received at least one dose of pasireotide LAR and had indication-specific baseline primary biochemical tumor marker levels >ULN. Responder analysis are reported only for indications with minimum of 6 patients. Patients with missing Month 6 assessment were considered as non-responders.
Measure: Number; unit: Participants
Groups:
- All PNETS (Gastrinoma): One of the 10 types of PNETs analyzed
Arm/Group | All PNETS (Gastrinoma)
Number analyzed (Participants) | 20
Participants
  Baseline | 8
  Month 6 | 5

5. Secondary Outcome: PiNETs: Number of Patients Attaining Normalization or a More Than 50% Reduction in Primary Biochemical Tumor Marker
Description: Specific primary biochemical tumor markers were used to assess the efficacy of pasireotide in PNETs. A Month 6 responder was defined as the patients who either attained normalization or greater than 50% reduction from baseline in the level of the primary biochemical tumor marker at Month 6.
Time Frame: Baseline, month 6
Population: as for outcome 4
Measure: Number; unit: Participants
Groups:
- All PiNETS (Prolactinoma): One of the 10 types of PiNETs analyzed
Arm/Group | All PiNETS (Prolactinoma)
Number analyzed (Participants) | 39
Participants
  Baseline | 7
  Month 6 | 9

6. Secondary Outcome: Nelson's Syndrome: Number of Patients Attaining Normalization or a More Than 50% Reduction in Primary Biochemical Tumor Marker
Description: Six patients with Nelson's syndrome met the responder's criteria of attaining normalization or a reduction of more than 50% in primary tumor marker at Month 6.
Time Frame: Baseline, month 6
Population: as for outcome 4
Measure: Number; unit: Participants
Groups:
- Nelson's Syndrome: Nelson's syndrome is associated with local tumor extension or invasion following a therapeutic bilateral adrenalectomy
Arm/Group | Nelson's Syndrome
Number analyzed (Participants) | 14
Participants
  Baseline | 6
  Month 6 | 6

ADVERSE EVENTS:
Groups:
- Pancreatic NETs (PNETs); Pituitary NETs (PiNETs); Ectopic ACTH-secrting Tumors (EAS): Patients received pasireotide LAR at 60 mg approximately once every 28 days for 6 months during the core treatment period and additional treatment cycles up to a total of 48 months during the extension phase.
- Nelsons Syndrome: Nelson's syndrome is based on disease specific primary biochemical tumor markers. Patients received pasireotide LAR at 60 mg approximately once every 28 days for 6 months during the core treatment period and additional treatment cycles up to a total of 48.
Arm/Group | Pancreatic NETs (PNETs) | Pituitary NETs (PiNETs) | Ectopic ACTH-secrting Tumors (EAS) | Nelsons Syndrome
Serious Adverse Events (participants affected / at risk) | 10/25 | 8/72 | 5/7 | 9/14
Other Adverse Events (participants affected / at risk) | 23/25 | 71/72 | 7/7 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pancreatic NETs (PNETs) (N=25) | Pituitary NETs (PiNETs) (N=72) | Ectopic ACTH-secrting Tumors (EAS) (N=7) | Nelsons Syndrome (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Haemophilia A without inhibitors (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Drug ineffective (General disorders) | 0 | 0 | 1 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pancreatic NETs (PNETs) (N=25) | Pituitary NETs (PiNETs) (N=72) | Ectopic ACTH-secrting Tumors (EAS) (N=7) | Nelsons Syndrome (N=14)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0
Palpitations (Cardiac disorders) | 2 | 1 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 8 | 0 | 3
Tachycardia (Cardiac disorders) | 3 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 3
Eustachian tube disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 0 | 1
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 0 | 2
Dry eye (Eye disorders) | 0 | 1 | 0 | 2
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 2
Photopsia (Eye disorders) | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 3 | 4 | 0 | 5
Visual acuity reduced (Eye disorders) | 0 | 3 | 0 | 2
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 8 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 11 | 2 | 5
Abdominal pain lower (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 9 | 2 | 7
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 6 | 1 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 43 | 3 | 11
Dry mouth (Gastrointestinal disorders) | 3 | 4 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 4 | 0 | 4
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 11 | 15 | 1 | 9
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 4 | 1 | 3
Asthenia (General disorders) | 4 | 10 | 0 | 2
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 1 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 10 | 1 | 7
Hypothermia (General disorders) | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 1 | 8 | 0 | 1
Injection site pruritus (General disorders) | 0 | 0 | 0 | 2
Injection site urticaria (General disorders) | 0 | 0 | 1 | 1
Local swelling (General disorders) | 2 | 0 | 0 | 1
Malaise (General disorders) | 1 | 4 | 0 | 0
Oedema peripheral (General disorders) | 5 | 1 | 1 | 0
Pyrexia (General disorders) | 2 | 4 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 3 | 17 | 0 | 3
Hepatic steatosis (Hepatobiliary disorders) | 0 | 9 | 0 | 0
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 2
Bone abscess (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 2
Cystitis (Infections and infestations) | 0 | 1 | 1 | 0
Ear infection (Infections and infestations) | 1 | 2 | 1 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Fungal oesophagitis (Infections and infestations) | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 4 | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 7 | 1 | 3
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 2
Tooth infection (Infections and infestations) | 1 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 8 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 7 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 2
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Inflammation of wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 0 | 1
Blood corticotrophin increased (Investigations) | 0 | 0 | 0 | 2
Blood glucagon decreased (Investigations) | 0 | 2 | 0 | 1
Blood glucose increased (Investigations) | 1 | 7 | 1 | 1
Blood insulin increased (Investigations) | 0 | 0 | 0 | 1
Body temperature fluctuation (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram QRS complex abnormal (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 2 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 2 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 5 | 1 | 2
Glycosylated haemoglobin increased (Investigations) | 2 | 4 | 0 | 2
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 1
Insulin-like growth factor decreased (Investigations) | 0 | 4 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 3 | 5 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 5 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 16 | 2 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 26 | 4 | 11
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0 | 3
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 1 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 4 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 8 | 0 | 3
Formication (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 5 | 11 | 2 | 4
Horner's syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1 | 0 | 2
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 1 | 0 | 2
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 3 | 1 | 0 | 2
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 1
Tremor (Nervous system disorders) | 1 | 1 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 7 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Polyuria (Renal and urinary disorders) | 2 | 1 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Hypomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 2 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 4 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Flushing (Vascular disorders) | 3 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 2 | 0 | 1
Hypertension (Vascular disorders) | 0 | 5 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Poor venous access (Vascular disorders) | 0 | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.